CLINICAL TRIAL: NCT03695003
Title: The Acute and Chronic Cognitive Effects of a Sage Extract: a Randomized, Placebo Controlled Study in Healthy Humans
Brief Title: Cognitive Effects of Sage in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Emma Wightman, Senior Lecturer, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 55C2
Record Dates: First submitted 2018-09-20; First posted 2018-10-03 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Cognitive Change; Mood Change
Keywords: Sage; Terpene; Polyphenol; Cognition; Mood

STUDY DESIGN:
Intervention Model Description: The study will follow a randomised, double-blind, placebo-controlled, parallel groups design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind. Randomized by a disinterested third party. Placebo and active capsules matched for aesthetics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 600 mg sage/polyphenol combination (Active Comparator): 600 mg of this sage/polyphenol combination will be consumed, via capsule, per day for 29 days.
  Interventions: Dietary Supplement: Cognivia
- Placebo (Placebo Comparator): The same number of aesthetically similar capsules will be consumed per day for 29 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cognivia — Cognivia is a trademarked sage/polyphenol combination dietary supplement from Nexira
  Arms: 600 mg sage/polyphenol combination
Dietary Supplement: Placebo — Placebo control capsules were prepared by Nexira also and are aesthetically identical to the Cognivia capsules
  Arms: Placebo

SUMMARY:
Extracts of sage and polyphenols have separately been reported to interact with central nervous system (CNS) mechanisms relevant to cognitive performance but, to date, no trial has combined these interventions. The current study investigates the effects of this combined intervention in N=90 healthy males and females between 30-60 yrs, at 600 mg versus placebo, on cognition and mood over a 29 day period.

DETAILED DESCRIPTION:
Improved cognitive performance has been observed in humans following supplementation of sage extracts; including recall and mental arithmetic ability. Aspects of mood have also shown improvements; e.g. increased alertness, calmness and contentedness and reduced mental fatigue. These effects are believed to be underpinned by interactions with cholinergic and GABA pathways. Polyphenols too have shown promise in boosting cognition and mood and interaction with vasodilatory pathways and GABA neurotransmission are purported to be the likely mechanisms involved. Research has yet to investigate if a combination of sage terpenes and polyphenols could be even more efficacious via synergistic interaction.The current study investigates the effects of a 600 mg sage/polyphenol combination on cognition and mood in N=90 healthy male and female participants between the ages of 30-60 yrs acutely; on day 1 of supplementation, and chronically; after 29 days. Cognitive and mood data will also be collected every 7 days in the interim via a mobile phone cognitive task battery.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health.
* Aged 30 to 60 years at the time of giving consent
* In daytime employment and/or higher education

Exclusion Criteria:

* Have any pre-existing medical condition/illness which will impact taking part in the study NOTE: the explicit exceptions to this are controlled (medicated) arthritis, asthma, hay fever, high cholesterol and reflux-related conditions. There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance.
* Are currently taking prescription medications NOTE: the explicit exceptions to this are contraceptive and hormone replacement treatments for female participants where symptoms are stable and treatment will not change during the course of the study, those medications used in the treatment of arthritis, high cholesterol and reflux-related conditions; and those taken 'as needed' in the treatment of asthma and hay fever. As above, there may be other instances of medication use which, where no interaction with the active treatments is likely, participants may be able to progress to screening.
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18.5-30 kg/m2
* Are pregnant, seeking to become pregnant or lactating
* Have learning and/or behavioural difficulties such as dyslexia or ADHD
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoker
* excessive caffeine intake (>500 mg per day)
* Have food intolerances/ sensitivities
* Have taken antibiotics, prebiotics or probiotics (including drinks. Eg. Yakult or Actimel) within the past 8 weeks
* Have any health condition that would prevent fulfillment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Sleep disturbances (including night-shift work) and/ or are taking sleep aid medication
* Any known active infections
* Does not have a bank account (required for payment)
* Are non-compliant with regards treatment consumption (see 4.3)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Acute change in global cognitive task performance | 120 minutes and 240 minutes post dose on day 1 of treatment supplementation
  Changes in executive function, working memory, spatial memory, secondary memory and attention as compared to pre-treatment performance on day 1. All tasks have the same x3 outcome measures; accuracy (% correct), errors (% incorrect) and speed (milliseconds) and the individual task scores will therefore be collapsed into global cognitive domains.
Acute changes in mood; as assessed by the Bond-Lader mood scales | 120 minutes and 240 minutes post dose on day 1 of treatment supplementation
  The Bond-Lader mood visual analogue scales will be used at baseline and 120- and 240-minutes post dose on day 1. The derived scores on alertness, calmness and contentedness will be 'changed-from-baseline' and this score compared across the treatments.
Interim changes in global cognitive task performance | Day 7, day 14, day 21 and day 28
  Changes in attention, executive function, working memory and episodic memory as compared to pre-treatment performance on day 1. All tasks have the same x3 outcome measures; accuracy (% correct), errors (% incorrect) and speed (milliseconds) and the individual task scores will therefore be collapsed into global cognitive domains.
Chronic changes in cognitive task performance | Pre-dose, 120 minutes and 240 minutes post-dose on day 29 of treatment supplementation
  Changes in executive function, working memory, spatial memory, secondary memory and attention as compared to pre-treatment performance on day 1. All tasks have the same x3 outcome measures; accuracy (% correct), errors (% incorrect) and speed (milliseconds) and the individual task scores will therefore be collapsed into global cognitive domains.
Chronic changes in mood; as assessed by the Bond-Lader mood scales | Pre-dose, 120 minutes and 240 minutes post dose on day 29 of treatment supplementation
  The Bond-Lader mood visual analogue scales will be used at baseline and 120- and 240-minutes post dose on day 29. The derived scores on alertness, calmness and contentedness will be 'changed-from-baseline' and this score compared across the treatments.
Change in prospective memory performance; as assessed by a prospective memory task (the prospective remembering video task) | Day 25 and day 29
  This individual task is called the Prospective Remembering Video Task (PRVP) and requires participants to remember a list of remembered locations and actions and identify these as they watch a video with them unfolding. The task is scored for difference in prospective memory/location learning performance between active and placebo on day 25 of supplementation period and also the difference in amount of memory decay of prospective memory/location learning on day 29 of treatment supplementation.
Acute changes in mood; as assessed by the 'state, trait anxiety inventory' (STAI) | 120 minutes and 240 minutes post dose on day 29 of treatment supplementation
  The STAI will be used at baseline and 120- and 240-minutes post dose on day 1. The anxiety scores will be 'changed-from-baseline' and this score compared across the treatments.
Chronic changes in mood; as assessed by the 'state, trait anxiety inventory' (STAI) | 120 minutes and 240 minutes post dose on day 29 of treatment supplementation
  The STAI will be used at baseline and 120- and 240-minutes post dose on day 29. The anxiety scores will be 'changed-from-baseline' and this score compared across the treatments.

SECONDARY OUTCOMES:
Acute changes in blood pressure | 120 minutes and 240 minutes post dose on day 1 of treatment supplementation
  Changes in blood pressure (BP) as compared to pre-dose BP on day 1. BP is assessed via forearm cuff and provides systolic and diastolic BP.
Chronic changes in blood pressure | Pre-dose, 120 minutes and 240 minutes post dose on day 29 of treatment supplementation
  Changes in blood pressure (BP) as compared to pre-dose BP on day 1. BP is assessed via forearm cuff and provides systolic and diastolic BP.
Acute changes in heart rate | 120 minutes and 240 minutes post dose on day 1 of treatment supplementation
  Changes in heart rate (HR) as compared to pre-dose HR on day 1. HR is assessed via forearm cuff.
Chronic changes in heart rate | Pre-dose, 120 minutes and 240 minutes post dose on day 29 of treatment supplementation
  Changes in heart rate (HR) as compared to pre-dose HR on day 1. HR is assessed via forearm cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Wightman, Dr, Principal Investigator — Northumbria University
Locations (1):
- Brain Performance and Nutrition Research Centre, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The IPD will be shared among the named investigators and Nexira only.

DOCUMENTS (1):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT03695003/Prot_000.pdf